CLINICAL TRIAL: NCT02191462
Title: A Randomized, Double-blind, Cross-over Study of the Pharmacokinetics of Three Dosages of Niagen in Healthy Subjects
Brief Title: A Study of the Pharmacokinetics of Three Dosages of Niagen in Healthy Subjects
Acronym: 14NBHC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KGK Science Inc. (Industry)
Collaborators: ChromaDex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 14NBHC
Record Dates: First submitted 2014-07-11; First posted 2014-07-16 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Pharmacokinetics
Keywords: Pharmacokinetics; Niagen; Nicotinamide riboside
MeSH Terms: interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Niagen 100mg (Experimental): 1 Niagen capsule (1 x 100 mg capsule) and 9 Placebo capsules
  Interventions: Dietary Supplement: Niagen 100mg
- Niagen 300mg (Experimental): 3 Niagen capsules (3 x 100mg capsule) and 7 Placebo capsules
  Interventions: Dietary Supplement: Niagen 300mg
- 1000mg Niagen (Experimental): 10 Niagen capsules (10 x 100mg capsule)
  Interventions: Dietary Supplement: Niagen 1000mg

INTERVENTIONS:
Dietary Supplement: Niagen 100mg
  Arms: Niagen 100mg
Dietary Supplement: Niagen 300mg
  Arms: Niagen 300mg
Dietary Supplement: Niagen 1000mg
  Arms: 1000mg Niagen

SUMMARY:
The purpose of this study in to analyse the way in which the body processes Niagen (nicotinamide riboside) in healthy people. Blood and urine samples from subjects who are given a dose of Niagen will be analyzed for metabolites over the 24 hours after taking the dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male or female age 30-55 years
* BMI 18.5-29.9 kg/m2
* If female, subject is not of child bearing potential, OR Females of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result.
* Healthy as determined by laboratory results and medical history
* Agrees to maintain current level of physical activity throughout the study
* Agrees to avoid vitamins and St. John's Wort for 30 days prior to enrollment and during the study
* Agrees to avoid nutritional yeast, whey proteins, energy drinks, dairy products, grapefruit and grapefruit juice and alcohol 7 days prior to enrollment and during study
* Has given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

* Women who are pregnant, breastfeeding, or planning to become pregnant during the course of the trial.
* Use of natural health products (NHPs)/dietary supplements within 7 days prior to randomization and during the course of the study.
* Use of vitamins or St. John's Wort in the last 30 days before the study enrollment,
* Use of natural health products containing Nicotinamide riboside within 7 days prior to randomization and during the course of the study
* Use of nutritional yeast, whey proteins, energy drinks, grapefruit and grapefruit juice, dairy products, alcohol for 7 days prior to the study
* Subjects who are smokers
* Subjects with blood pressure ≥140/90
* Use of blood pressure medications
* Use of cholesterol lowering medications
* Metabolic diseases or chronic diseases
* Use of acute over the counter medication within 72 hours of test product dosing
* Unstable medical conditions as determined by the Qualified Investigator
* Immunocompromised individuals such as subjects that have undergone organ transplantation or subjects diagnosed with human immunodeficiency virus (HIV)
* Clinically significant abnormal lab results at screening (e.g. AST and/or ALT > 2 x ULN, and/or bilirubin > 2 x ULN) will be assessed by the Medical Investigator
* Subjects who have planned surgery during the course of the trial
* History of or current diagnosis of any cancer (except for successfully treated basal cell carcinoma) diagnosed less than 5 years prior to screening. Subjects with cancer in full remission more than 5 years after diagnosis are acceptable
* History of blood/bleeding disorders
* Blood donation in the past 2 months
* Alcohol abuse (>2 standard alcoholic drinks per day) or drug abuse within the past 6 months
* Participation in a clinical research trial within 30 days prior to randomization
* Allergy or sensitivity to study supplement ingredients or to any food or beverage provided during the study
* Individuals who are cognitively impaired and/or who are unable to give informed consent.
* Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
t1/2 (terminal half-life) | 24 hours
  24 hour dosing period; 3 dosing periods each separated by 7 day washout

OTHER OUTCOMES:
Area under the curve (AUC(0-24h) | 24 hours
  24 hour dosing period; 3 dosing periods each separated by 7 day washout
AUCI (AUC to infinity) | 24 hours
  24 hour dosing period; 3 dosing periods each separated by 7 day washout
AUC(0-24h)/AUCI | 24 hours
  24 hour dosing period; 3 dosing periods each separated by 7 day washout
Maximum observed concentration (Cmax) | 24 hours
  24 hour dosing period; 3 dosing periods each separated by 7 day washout
Time of maximum concentration (Tmax), | 24 hours
  24 hour dosing period; 3 dosing periods each separated by 7 day washout
λ (terminal disposition rate constant) | 24 hours
  24 hour dosing period; 3 dosing periods each separated by 7 day washout
AUCReftmax (Area under the curve to tmax) | 24 hours
  24 hour dosing period; 3 dosing periods each separated by 7 day washout
Blood Safety parameters | 24 hour dosing period; pre dose and 24 hr post dose
  CBC
Blood Safety parameters | 24 hour dosing period; pre dose and 24 hr post dose
  electrolytes
Blood Safety parameters | 24 hour dosing period; pre dose and 24 hr post dose
  glucose
Blood Safety parameters | 24 hour dosing period; pre dose and 24 hr post dose
  creatinine
Blood Safety parameters | 24 hour dosing period; pre dose and 24 hr post dose
  AST
Blood Safety parameters | 24 hour dosing period; pre dose and 24 hr post dose
  ALT
Blood Safety parameters | 24 hour dosing period; pre dose and 24 hr post dose
  GGT
Blood Safety parameters | 24 hour dosing period; pre dose and 24 hr post dose
  uric acid
Blood Safety parameters | 24 hour dosing period; pre dose and 24 hr post dose
  bilirubin
Vital Signs | 24 hour period: pre-dose, 1h, 4h, 6h, 12h, 24h post-dose
  Heart Rate
Vital Signs | 24 hour period: pre-dose, 1h, 4h, 6h, 12h, 24h post-dose
  Blood Pressure

CONTACTS AND LOCATIONS:
Overall Officials: Dale Wilson, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Synergize Inc., London, Ontario, Canada